CLINICAL TRIAL: NCT06742372
Title: Effects of Combined Exercise Training Modality on Diaphragm Function and Performance
Brief Title: Effects of Combined Exercise Training Modality
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Zeliha ÇELİK, Asst. Prof., Amasya University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 310783
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Healthy Individuals (Controls)

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combined inspiratory and aerobic exercise training (Experimental)
  Interventions: Other: combined inspiratory and aerobic exercise training
- aerobic exercise training (Experimental)
  Interventions: Other: aerobic exercise training

INTERVENTIONS:
Other: combined inspiratory and aerobic exercise training — combined inspiratory and aerobic exercise training will be performed in healthy individuals
  Arms: combined inspiratory and aerobic exercise training
Other: aerobic exercise training — aerobic exercise training will be performed in healthy individuals
  Arms: aerobic exercise training

SUMMARY:
This study aims to investigate the effects of combined Inspiratory Muscle Training and aerobic exercise on diaphragm and pulmonary functions, respiratory muscle function, performance, and body composition

ELIGIBILITY:
Inclusion Criteria:aged between 18 and 40 years who have physical activity levels above 600 MET-min/week -

Exclusion Criteria:Individuals who were diagnosed with any cardiopulmonary or other chronic diseases, have any infections or limitations preventing them from doing an activity during assessment or intervention, do exercise regularly, and have smoked over 10 pack-years

-

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Respiratory muscle strength | First day
  Maximal inspiratory and expiratory muscle strength will be evaluated using mouth pressure device .
diaphragm thickness | Second day
diaphragm stiffness | Second day

SECONDARY OUTCOMES:
Inspiratory muscle endurance | First day
FEV1 | First day
FVC | First day
FEV1/FVC | First day
PEF | First day
FEF2575 | First day
Running Based Anaerobic Sprint Test (RAST test) | Second day

CONTACTS AND LOCATIONS:
Locations (1):
- Amasya University, Amasya, Turkey (Türkiye)

REFERENCES:
- [Derived] Celik Z, Guzel NA, Allahverdiyeva S, Sendur HN, Cerit MN. Effects of simultaneous aerobic and inspiratory muscle training on diaphragm function, respiratory muscle strength, endurance, and fatigue index: randomized-controlled trial. Eur J Appl Physiol. 2025 Dec;125(12):3769-3783. doi: 10.1007/s00421-025-05868-1. Epub 2025 Jul 2. PMID 40601012